CLINICAL TRIAL: NCT00518609
Title: Prevention of Infection in Indian Neonates - Phase I Observational Study
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); All India Institute of Medical Sciences (Other); TN Medical College, Mumbai (Other); Department of Health and Family Welfare, Orissa (Other); SCB Medical College, Cuttack (Other); Capital Hospital, Bhubaneswar (Other); Ispat General Hospital, Rourkela (Other); Kalinga Hospital, Bhubaneswar (Other); University of Maryland (Other)
Responsible Party: Sponsor
Other Study IDs: GN 07 Phase I; U01HD040574 (NIH); NCT00098176 (obsolete NCT alias)
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Sepsis
Keywords: Neonatal; Sepsis; Global Network; Antibiotics; India; International; Maternal and child health
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Indian Neonates: All hospitalized neonates (all live born infants <60 days of age, independent of birth weight and gestational age) brought to hospital, with the diagnosis of suspected sepsis.

SUMMARY:
India, with one of the world's largest populations, continues to struggle with extremely high infant and neonatal mortality rates. Neonatal infection (sepsis) now accounts for 50 percent of deaths among community-born (and 20 percent of mortality among hospital-born) infants. This study is the first phase of a multi-phase project investigating interventions to prevent neonatal infection in India.

DETAILED DESCRIPTION:
Invasive bacterial infections encompass clinical diagnoses of septicemia, pneumonia, and meningitis. Together, these infections are termed "neonatal sepsis" and account for over half of the newborn deaths at the district and sub-district level in India. Sepsis is the most common (80-90 percent) primary diagnosis for admission in Indian hospitals. Phase 1 of this study is a prospective, epidemiologic study involving over 1,000 community-based and hospital populations of newborn infants. It includes identifying all infants born in study hospitals and those brought to the hospitals with suspected sepsis; obtaining blood cultures from these infants and identifying the sepsis-causing bacteria; screening of all bacterial strains isolated from blood cultures for antimicrobial resistance; collecting basic demographic, risk factor, and treatment data on each case; and developing a computer-based system/network for data management. A village-level surveillance system was put in place to identify women during their pregnancy; monitor pregnancy outcomes; and establish a mechanism for referral of all potentially septic infants to participating clinics or hospitals for evaluation, including the collection of blood cultures. Potential sources of bacteria causing sepsis will be identified using molecular epidemiologic techniques. This involves matching septic infants' blood isolates with other colonizing isolates obtained from screening skin, throat, and stool cultures in the infant and skin and vaginal cultures from their mothers.

ELIGIBILITY:
Inclusion Criteria:

* Age <60 days
* A diagnosis of suspected sepsis/pneumonia, based on the presence of at least one of the following symptoms at admission: poor feeding/poor sucking, decreased activity/lethargy, fever, hypothermia, cyanosis, diarrhea, abdominal distension, seizures, apneic spells, sclerema, bleeding, jaundice, tachypnea, chest wall retractions, shock.
* Born in one of the participating hospitals or in village inside catchment area If the screening physician does not suspect sepsis, even in the presence of one or more of the above signs, the baby should not be enrolled.

Exclusion Criteria:

• The presence of major congenital anomalies A major congenital anomaly is defined as any malformation that is felt to be life-threatening or that requires surgical intervention. If the medical officer is uncertain whether an anomaly is life-threatening, he/she should not enroll the infant.

Max Age: 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1326 (Actual)
Dates: Start 2003-07; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pinaki Panigrahi, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (3):
- India (3):
  - Capital Hospital, Bhubaneswar, Odisha
  - Kalinga Hospital, Bhubaneswar, Odisha
  - Ispat General Hospital, Rourkela, Odisha

REFERENCES:
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: RTI International — http://www.rti.org